CLINICAL TRIAL: NCT00648245
Title: A Phase 2a, Double Blind, Placebo Controlled, Multicenter, Dose Escalation Study to Evaluate the Safety and Efficacy of BIO 11006 Inhalation Solution in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Effectiveness and Safety of BIO-11006 Inhalation Solution to Treat the Overproduction of Mucus and Inflammation in COPD
Acronym: BREATH-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarck Pharmaceuticals, Ltd. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Ted Murphy, BioMarck Pharmaceuticals, Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIM-CL-003; 5R44HL073591 (NIH)
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; Chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: BIO-11006 Inhalation Solution
- 2 (Experimental)
  Interventions: Drug: BIO-11006 Inhalation Solution
- 3 (Experimental)
  Interventions: Drug: BIO-11006 Inhalation Solution
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- 5 (Experimental)
  Interventions: Drug: BIO-11006

INTERVENTIONS:
Drug: BIO-11006 Inhalation Solution — 75 mg of BIO-11006 administered once per day for 21 days by nebulizer
  Arms: 1
Drug: BIO-11006 Inhalation Solution — 150 mg of BIO-11006 administered once per day for 21 days by nebulizer
  Arms: 2
Drug: BIO-11006 Inhalation Solution — 75 mg of BIO-11006 administered twice per day for 21 days by nebulizer
  Arms: 3
Drug: Placebo — Placebo given once daily for 21 days by nebulizer
  Arms: 4
Drug: BIO-11006 — 125 mg BIO-11006 given twice per day for 21 days by nebulizer
  Arms: 5

SUMMARY:
The symptoms associated with COPD include overproduction of mucus and inflammation in the lungs. Overproduction of mucus results in impaired lung function and it encourages bacterial growth and associated COPD exacerbations. Therefore, a treatment that inhibits mucus overproduction or blocks inflammation could benefit COPD patients. The drug under evaluation in this study, BIO-11006 Inhalation Solution, is a new drug that may inhibit overproduction of mucus and may have important anti-inflammatory properties.

DETAILED DESCRIPTION:
COPD encompasses a number of chronic lung disorders that obstruct the airways and may be accompanied by airway hyperactivity. The most common form of COPD is a combination of chronic bronchitis and emphysema. Many of the signs and symptoms associated with chronic bronchitis are a result of airway mucus hypersecretion induced by chronic inflammation of the airways. Clinically, mucus hypersecretion results in impaired gas exchange and compromised mucociliary clearance, encouraging bacterial colonization and associated exacerbations. A treatment that inhibits mucus hypersecretion or blocks inflammation could benefit COPD patients with chronic bronchitis. The drug under evaluation in this study, BIO 11006, is a new therapeutic agent that may inhibit mucus secretion and may have important anti inflammatory properties. In this study, BIO-11006 will be administered to COPD patients with chronic bronchitis, and the effects lung function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable male or female outpatients, 45 years of age or older
* Active COPD with chronic bronchitis indicated by: (1) FEV1 = 40% to 70%, (2) FEV1/FVC ≤70%, (3)Chronic productive cough for 3 months in each of 2 successive years, and (4) Sputum (phlegm) production at least several days a week over the past 4 weeks
* Current or previous smoker with a 20-pack year history

Exclusion Criteria:

* Treatment with oral prednisone during the 6 weeks before enrollment
* Changed inhaled corticosteroid dose or long acting bronchodilator dose during the 6 weeks before enrollment
* Treatment with oxygen (with the exception of night time oxygen) during the 6 weeks before enrollment
* Current asthma as determined by the investigator
* Change in smoking status during the previous 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety of BIO-11006 when administered once or twice daily for 21 days to subjects with COPD by assessing adverse events, physical exams, vital signs, pulmonary function, 12 lead electrocardiogram, clinical blood chemistries, hematology, and urinalysis. | Throughout study

SECONDARY OUTCOMES:
Efficacy of BIO-11006 when administered once or twice daily for 21 days to subjects with COPD by assessing the change from baseline in pulmonary function. | Day 21 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ted C Murphy, Ph.D, Study Director — BioMarck Pharmaceuticals, Ltd.
Locations (14):
- United States (14):
  - Pulmonary Associates, Glendale, Arizona
  - Greater Los Angeles Healthcare System, Los Angeles, California
  - Bay Pines VA Heatlhcare System, Bay Pines, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Southeastern Lung Care, Decatur, Georgia
  - University of Louisville, Louisville, Kentucky
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Southeastern Research Center, LLC, Winston-Salem, North Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VAMC, Houston, Texas
  - Diagnostics Research Group, San Antonio, Texas

REFERENCES:
- See also: Click here for more information about the sponsor of this study — http://www.biomarck.com